CLINICAL TRIAL: NCT00805766
Title: Clinical Study to Assess the Efficacy and Safety of Increased Dose of TA-650 in Patients With Crohn's Disease (CD)
Brief Title: Efficacy and Safety of Increased Dose of TA-650 (Infliximab) in Patients With Crohn's Disease (CD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA-650-19
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Results first posted 2012-12-05 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Crohn's Disease
Keywords: Infliximab; REMICADE; Crohn's disease
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TA-650 (Experimental)
  Interventions: Drug: TA-650

INTERVENTIONS:
Drug: TA-650 — (1) Screening Period: 5 mg/kg of TA-650 will be intravenously infused over a period of more than 2 hours at week 0. If patients do not meet the Eligibility Criteria at week 8, they will be administered 5 mg/kg of TA-650 at week 8. (2) Increased Dose Period: 10 mg/kg of TA-650 will be intravenously infused over a period of more than 2 hours every 8 weeks for 32 weeks.
  Other Names: Infliximab

SUMMARY:
The purpose of this study is to assess the efficacy, safety and pharmacokinetics after administration of 10mg/kg TA-650 every 8 weeks to patients with Crohn's disease showing an insufficient response to previous treatment with 5 mg/kg of REMICADE every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Crohn's disease
* Patients who have relapsed with symptoms associated with Crohn's disease within 8 weeks in spite of maintenance treatment with 5mg/kg REMICADE every 8 weeks, and who are judged to be showing an insufficient response to the previous treatment by their physician

Exclusion Criteria:

* Severe intestinal strictures (which may have an effect on the number of loose stools or diarrhea or dilation of the colon or small bowel proximal to the stricture on barium radiograph or an inability to traverse the stricture at endoscopy), a diagnosis of short bowel syndrome, or previous stoma surgery
* The presence of significant internal fistula (possibility that surgery might be needed, etc.) is confirmed
* A history of a serious infusion reaction to REMICADE
* Pregnant, lactating, and probably pregnant women
* Patients who have participated in other trials and have been administered other investigational products within 12 weeks before consent
* Patients judged to be inadequate to participate in this study by their physician

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toshifumi Hibi, Professor, Study Chair — Department of Internal Medicine, Keio University School of Medicine
Locations (4):
- Japan (4):
  - Investigational site, Hokkaido
  - Investigational site, Kansai
  - Investigational site, Kanto
  - Investigational site, Kyushu

RESULTS

PARTICIPANT FLOW:
Groups:
- TA-650: Screening period: From the beginning of TA-650 5 mg/kg administration to the beginning of TA-650 10 mg/kg administration in the increased dose period in order to confirm that the effects of treatment with TA-650 5 mg/kg at 8-week intervals were insufficient. The screening period was to be up to 16 weeks. Patients who did not satisfy the dose-increasing criteria discontinued study treatment.Patients who discontinued study treatment during the screening period were to be evaluated until withdrawal.
  Increased dose period: From the beginning of administration of TA-650 10 mg/kg to evaluation at week 40. Patients who discontinued study treatment during the increased dose period were to be evaluated until withdrawal.
Period: Screening Period
Arm/Group | TA-650
Started | 45
Completed | 39
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 2
Not completed — Pregnancy | 1
Not completed — Responder | 2
Period: Increased Dose Period
Arm/Group | TA-650
Started | 39
Completed | 26
Not Completed | 13
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 7
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | TA-650
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] — Screening period:
  years | 29.5 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Screening period:
  Participants
    Female | 14
    Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Median Crohn's Disease Activity Index (CDAI) Change From Week 0 to Week 8 in the Increased Dose Period
Description: To confirm the decrease in median CDAI at week 8 by ≥ 50 points compared to the CDAI score at week 0 in the increased dose period. In the indication of CDAI change, decrease in CDAI was expressed by positive numbers. CDAI is a research tool used to quantify the symptoms of patients with Crohn's disease. CDAI scores generally range from 0 to 600 points. Clinical remission = CDAI < 150 points. Moderate disease = CDAI 220 - 450 points. Severe disease = CDAI > 450 points.
Time Frame: Increased Dose Period (Week 0 to Week 8)
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | TA-650
Number analyzed (Participants) | 33
units on a scale | 95.0 [70.0 to 134.0]

2. Secondary Outcome: CDAI at Each Evaluation Time Point in the Increased Dose Period
Description: CDAI is a research tool used to quantify the symptoms of patients with Crohn's disease. CDAI scores generally range from 0 to 600 points. Clinical remission = CDAI < 150 points. Moderate disease = CDAI 220 - 450 points. Severe disease = CDAI > 450 points.
Time Frame: Increased Dose Period (every 4 weeks for up to 40 weeks)
Population: One patient whose data after week 4 in the increased dose period was missing was excluded from the analysis. Patients whose the outcome measure were not assessed at a time point due to dropout were excluded from the analysis of the time point.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | TA-650
Number analyzed (Participants) | 38
units on a scale
  Week 0 | 296.5 [185 to 523]
  Week 4: number analyzed (Participants) | 37
  Week 4 | 119.0 [17 to 318]
  Week 8: number analyzed (Participants) | 33
  Week 8 | 194.0 [51 to 456]
  Week 12: number analyzed (Participants) | 30
  Week 12 | 126.0 [14 to 419]
  Week 16: number analyzed (Participants) | 29
  Week 16 | 182.0 [70 to 398]
  Week 20: number analyzed (Participants) | 29
  Week 20 | 121.0 [13 to 304]
  Week 24: number analyzed (Participants) | 28
  Week 24 | 197.5 [81 to 379]
  Week 28: number analyzed (Participants) | 28
  Week 28 | 105.0 [4 to 289]
  Week 32: number analyzed (Participants) | 27
  Week 32 | 163.0 [72 to 410]
  Week 36: number analyzed (Participants) | 27
  Week 36 | 141.0 [-3 to 315]
  Week 40: number analyzed (Participants) | 26
  Week 40 | 148.5 [41 to 407]
  Week 40 (the last time point) | 210.5 [34 to 479]

3. Secondary Outcome: CDAI Remission Rates at Each Evaluation Time Point in the Increased Dose Period
Description: as for outcome 2
Time Frame: Increased Dose Period (every 4 weeks for up to 40 weeks)
Population: Patients whose the outcome measure were not assessed at a time point due to dropout were excluded from the analysis of the time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TA-650
Number analyzed (Participants) | 39
percentage of participants
  Week 4: number analyzed (Participants) | 37
  Week 4 | 59.5 [42.1 to 75.2]
  Week 8: number analyzed (Participants) | 33
  Week 8 | 39.4 [22.9 to 57.9]
  Week 12: number analyzed (Participants) | 30
  Week 12 | 70.0 [50.6 to 85.3]
  Week 16: number analyzed (Participants) | 29
  Week 16 | 31.0 [15.3 to 50.8]
  Week 20: number analyzed (Participants) | 29
  Week 20 | 58.6 [38.9 to 76.5]
  Week 24: number analyzed (Participants) | 28
  Week 24 | 28.6 [13.2 to 48.7]
  Week 28: number analyzed (Participants) | 28
  Week 28 | 60.7 [40.6 to 78.5]
  Week 32: number analyzed (Participants) | 27
  Week 32 | 37.0 [19.4 to 57.6]
  Week 36: number analyzed (Participants) | 27
  Week 36 | 59.3 [38.8 to 77.6]
  Week 40: number analyzed (Participants) | 26
  Week 40 | 50.0 [29.9 to 70.1]
  Week 40 (the last time point) | 41.0 [25.6 to 57.9]

4. Secondary Outcome: CDAI Change at Each Evaluation Time Point in the Increased Dose Period
Description: as for outcome 1
Time Frame: Increased Dose Period (every 4 weeks for up to 40 weeks)
Population: as for outcome 2
Measure: Median (Full Range); unit: units on a scale
Arm/Group | TA-650
Number analyzed (Participants) | 38
units on a scale
  Week 0 to Week 4: number analyzed (Participants) | 37
  Week 0 to Week 4 | 163.0 [24 to 356]
  Week 0 to Week 8: number analyzed (Participants) | 33
  Week 0 to Week 8 | 95.0 [-26 to 301]
  Week 0 to Week 12: number analyzed (Participants) | 30
  Week 0 to Week 12 | 161.0 [-17 to 342]
  Week 0 to Week 16: number analyzed (Participants) | 29
  Week 0 to Week 16 | 95.0 [-36 to 240]
  Week 0 to Week 20: number analyzed (Participants) | 29
  Week 0 to Week 20 | 164.0 [-63 to 343]
  Week 0 to Week 24: number analyzed (Participants) | 28
  Week 0 to Week 24 | 100.0 [-21 to 252]
  Week 0 to Week 28: number analyzed (Participants) | 28
  Week 0 to Week 28 | 156.5 [0 to 352]
  Week 0 to Week 32: number analyzed (Participants) | 27
  Week 0 to Week 32 | 110.0 [-28 to 279]
  Week 0 to Week 36: number analyzed (Participants) | 27
  Week 0 to Week 36 | 139.0 [20 to 359]
  Week 0 to Week 40: number analyzed (Participants) | 26
  Week 0 to Week 40 | 95.0 [-54 to 390]
  Week 0 to 40(last measurable time point) | 87.0 [-63 to 390]

5. Secondary Outcome: Serum Concentration of TA-650 at Each Time Point
Time Frame: Screening Period (every 4 weeks for up to 16 weeks), Increased Dose Period (every 4 weeks for up to 40 weeks), a total of 56 weeks
Population: as for outcome 3
Measure: Median (Full Range); unit: μg/mL
Arm/Group | TA-650
Number analyzed (Participants) | 39
μg/mL
  Screening Period (SP), Week 0 (pre-dose) | 1.12 [0.00 to 13.29]
  SP, 1 hr after treatment end for week 0 | 97.74 [42.98 to 132.99]
  SP, Week 4 | 4.93 [0.00 to 27.70]
  SP, Week 8 | 0.30 [0.00 to 10.69]
  SP, Week 12: number analyzed (Participants) | 2
  SP, Week 12 | 5.25 [0.00 to 10.49]
  SP, Week 16: number analyzed (Participants) | 2
  SP, Week 16 | 0.79 [0.00 to 1.57]
  Increased dose Period(IP), Week0 (pre-dose) | 0.30 [0.00 to 10.69]
  IP, 1 hr after treatment end for week 0 | 191.24 [144.56 to 293.32]
  IP, Week 4: number analyzed (Participants) | 37
  IP, Week 4 | 9.93 [0.00 to 43.55]
  IP, Week 8: number analyzed (Participants) | 33
  IP, Week 8 | 1.29 [0.00 to 21.82]
  IP, Week 12: number analyzed (Participants) | 31
  IP, Week 12 | 11.20 [0.00 to 48.30]
  IP, Week 16 (pre-dose): number analyzed (Participants) | 29
  IP, Week 16 (pre-dose) | 1.31 [0.00 to 23.67]
  IP, 1hr after administration at week 16: number analyzed (Participants) | 29
  IP, 1hr after administration at week 16 | 203.16 [140.33 to 306.48]
  IP, Week 20: number analyzed (Participants) | 29
  IP, Week 20 | 8.71 [0.00 to 44.62]
  IP, Week 24: number analyzed (Participants) | 28
  IP, Week 24 | 1.83 [0.00 to 25.84]
  IP, Week 28: number analyzed (Participants) | 28
  IP, Week 28 | 9.97 [0.00 to 43.55]
  IP, Week 32: number analyzed (Participants) | 27
  IP, Week 32 | 1.60 [0.00 to 23.11]
  IP, Week 36: number analyzed (Participants) | 27
  IP, Week 36 | 12.72 [0.00 to 54.37]
  IP, Week 40: number analyzed (Participants) | 26
  IP, Week 40 | 2.18 [0.00 to 22.60]

6. Secondary Outcome: Antibody to TA-650 Determination
Time Frame: Screening Period (Week 0 to Week 16), Increased Dose Period (Week 0 to Week 40)
Measure: Number; unit: percentage of participants
Arm/Group | Screening Period | Increased Dose Period
Number analyzed (Participants) | 39 | 39
percentage of participants
  Negative | 23.1 | 17.9
  Positive | 5.1 | 5.1
  Inconclusive | 71.8 | 76.9

ADVERSE EVENTS:
Groups:
- Entire Evaluation Period: Screening Period + Increased Dose Period
Arm/Group | Entire Evaluation Period | Screening Period | Increased Dose Period
Serious Adverse Events (participants affected / at risk) | 9/45 | 2/45 | 8/39
Other Adverse Events (participants affected / at risk) | 37/45 | 25/45 | 29/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Entire Evaluation Period (N=45) | Screening Period (N=45) | Increased Dose Period (N=39)
Crohn's disease (Gastrointestinal disorders) | 6 | 1 | 5
Melaena (Gastrointestinal disorders) | 1 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Entire Evaluation Period (N=45) | Screening Period (N=45) | Increased Dose Period (N=39)
Nasopharyngitis (Infections and infestations) | 12 | 3 | 11
Influenza (Infections and infestations) | 3 | 1 | 2
Gastroenteritis (Infections and infestations) | 2 | 0 | 2
Pharyngitis (Infections and infestations) | 2 | 0 | 2
Bronchitis (Infections and infestations) | 1 | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 1
Otitis externa (Infections and infestations) | 1 | 1 | 0
Otitis media (Infections and infestations) | 1 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 1
Anal fistula infection (Infections and infestations) | 1 | 1 | 0
DNA antibody positive (Investigations) | 18 | 15 | 4
Blood urine present (Investigations) | 2 | 2 | 1
Liver function test abnormal (Investigations) | 2 | 0 | 2
Protein urine present (Investigations) | 2 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Chest X-ray abnormal (Investigations) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 3 | 2 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 3 | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Polymorphic light eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1
Hot flush (Vascular disorders) | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Periodontitis (Gastrointestinal disorders) | 1 | 0 | 1
Renal mass (Renal and urinary disorders) | 1 | 0 | 1
Haematospermia (Reproductive system and breast disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other